CLINICAL TRIAL: NCT01320358
Title: A 3-month, Exploratory, Non-randomized, Multi-center, Open Label Study to Evaluate the Reliability, Safety and Usability of the Transplantation Sensor System Combined With Myfortic® in Adult Kidney Transplant Patients
Brief Title: Reliability, Safety and Usability of the Transplantation Sensor System Combined With Myfortic® in Adult Kidney Transplant Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Proteus Digital Health, Inc. (Industry); Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CPRO400A2201
Record Dates: First submitted 2011-03-21; First posted 2011-03-22 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Detection Accuracy; Patient Compliance
Keywords: Patient compliance; ECMPS-IEM; transplantation; renal maintenance; Proteus
MeSH Terms: conditions — Patient Compliance; Proteus Infections

ARMS (1):
- ECMPS-IEM (Experimental)
  Interventions: Drug: ECMPS-IEM

INTERVENTIONS:
Drug: ECMPS-IEM — ECMPS-IEM

SUMMARY:
The main purpose of this exploratory trial is to evaluate the reliability, safety and usability of the Transplantation Sensor System when the Ingestible Event Marker (IEM) is given in combination with ECMPS 360 mg tablets in adult renal transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 6 months post-transplantation and in stable clinical condition
* Treatment with ECMPS doses between 720 mg/day and 1440 mg/day or MMF doses between1000 mg/day and 2000 mg/day, divided in two equal doses 12 hours apart and with no dose titrations planned for the duration of the trial
* Ability to independently take medication
* Successfully ingest a Placebo-IEM capsule with no difficulty

Exclusion Criteria:

* Inability to use the mobile phone provided for use in the clinical trial
* Any episodes of acute rejection in the previous 3 months
* Presence of cognitive impairment
* Active alcohol or drug abuse
* History of dysphagia, or inflammatory bowel disease, or gastrointestinal conditions or surgery that has modified the normal luminal flow of the gastrointestinal tract (e.g. Whipple procedure, bariatric surgery or Roux-en-Y)
* Known allergies, including history of skin reactions to patches, that could preclude safe participation in the study Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-05-10 (Actual); Primary Completion 2011-11-18 (Actual); Study Completion 2011-11-18 (Actual)

PRIMARY OUTCOMES:
To assess the reliability of the Raisin technology defined as accuracy and precision in detecting directly observed ingestion of ECMPS-IEM and Placebo-IEM. | 12 weeks

SECONDARY OUTCOMES:
the adherence (taking and scheduling) to prescribed ECMPS-IEM schedule with and without active feedback for two consecutive periods of 8 and 4 weeks each. | 12 weeks
the incidence and severity of adverse events observed during the utilization of the ECMPS-IEM and Proteus Personal Monitor (patch). | 12 weeks
the satisfaction and usability of the TSS by patients | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- Switzerland (5):
  - Kantonspital Aarau AG / Nephrologie, Aarau
  - University Hospital Basel, Basel
  - Inselspital Bern / Nephrology, Bern
  - Stadtspital Waid Zurich, Zurich
  - University Hospital Zurich, Zurich

REFERENCES:
- [Background] Fine RN, Becker Y, De Geest S, Eisen H, Ettenger R, Evans R, Rudow DL, McKay D, Neu A, Nevins T, Reyes J, Wray J, Dobbels F. Nonadherence consensus conference summary report. Am J Transplant. 2009 Jan;9(1):35-41. doi: 10.1111/j.1600-6143.2008.02495.x. PMID 19133930
- [Result] Eisenberger U, Wuthrich RP, Bock A, Ambuhl P, Steiger J, Intondi A, Kuranoff S, Maier T, Green D, DiCarlo L, Feutren G, De Geest S. Medication adherence assessment: high accuracy of the new Ingestible Sensor System in kidney transplants. Transplantation. 2013 Aug 15;96(3):245-50. doi: 10.1097/TP.0b013e31829b7571. PMID 23823651